CLINICAL TRIAL: NCT05375331
Title: Clinical and Genetic Markers of Bone Metabolism in Children Under One Year of Age in the Kazakh Population
Brief Title: Clinical and Genetic Markers of Bone Metabolism in Children Under One Year
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West Kazakhstan Medical University (Other)
Responsible Party: Principal Investigator, Irina Kim, Principal investigator of Department of Children's diseases, West Kazakhstan Medical University
Other Study IDs: 777.04.12.2020
Record Dates: First submitted 2022-04-24; First posted 2022-05-16 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Bone Remodeling Disorder; Child Development; Genetic Change

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study of children under one year of age for molecular genetic testing-VDR (rs1544410, rs2228570), RANKL (rs9594738, rs9594759) with the study of the frequency distribution of alleles and genotypes by polymorphisms, analysis of the relationship of molecular genetic markers with indicators of bone metabolism.

DETAILED DESCRIPTION:
Children under the age of one year of Kazakh nationality born in Aktobe will be examined.

Each child included in the study will have an individual registration card, where information about the health status of the child and the health status of the mother during pregnancy will be filled in.

A biochemical analysis will be determined for the level of calcium, phosphorus, calcitonin, parathyroid hormone, osteocalcin, vitamin D in blood serum and deoxypyridinoline in urine.

Blood will be taken to determine the genetic polymorphism of VDR (rs1544410, rs2228570), RANKL (rs9594738, rs9594759).

The state of bone tissue remodeling (osteocalcin, vitamin D, Ca, P, calcitonin, deoxypyridinoline) will be revealed The frequencies of allelic variants of the VDR (rs1544410, rs2228570), RANKL (rs9594738, rs9594759) genes in children under the age of one year in the population of Kazakhstan were determined.

ELIGIBILITY:
Inclusion Criteria:

-Children 0 -12 months old

Exclusion Criteria:

* Musculoskeletal system diseases;
* Severe chronic somatic diseases;
* Supplementation of vitamin D in a therapeutic dose;
* Lack of consent of the parents or legal representatives to participate in the study.

Ages: 1 Day to 1 Year | Sex: All
Age Groups: Child
Study Population: In accordance with the goal and objectives of the project, 245 children under the age of one year from the Kazakh population born in Aktobe will be examined. (N*-13500, p=16% n=204 +20%(41)=245 children).
  *N is the total fertility of children; n is how many children should be taken + 20% losses. total for research you need 245
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Optimization of the method for diagnosing bone metabolism disorders in children under one year old in the Kazakh population | 2 years
  The state of bone metabolism was assessed using the quantitative content of calcium, phosphorus, vitamin D, osteocalcin, and parathyroid hormone.

CONTACTS AND LOCATIONS:
Locations (1):
- Irina Kim, Aktobe, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bizzaro G, Antico A, Fortunato A, Bizzaro N. Vitamin D and Autoimmune Diseases: Is Vitamin D Receptor (VDR) Polymorphism the Culprit? Isr Med Assoc J. 2017 Jul;19(7):438-443. PMID 28786260
- [Result] Bao L, Chen M, Lei Y, Zhou Z, Shen H, Le F. Association between vitamin D receptor BsmI polymorphism and bone mineral density in pediatric patients: A meta-analysis and systematic review of observational studies. Medicine (Baltimore). 2017 Apr;96(17):e6718. doi: 10.1097/MD.0000000000006718. PMID 28445285
- [Result] Basit S. Vitamin D in health and disease: a literature review. Br J Biomed Sci. 2013;70(4):161-72. doi: 10.1080/09674845.2013.11669951. PMID 24400428
- [Result] Antonucci R, Locci C, Clemente MG, Chicconi E, Antonucci L. Vitamin D deficiency in childhood: old lessons and current challenges. J Pediatr Endocrinol Metab. 2018 Mar 28;31(3):247-260. doi: 10.1515/jpem-2017-0391. PMID 29397388